CLINICAL TRIAL: NCT01476384
Title: Postprandial Insulin Release and the Impact on Muscle Perfusion
Brief Title: Orthogonal Polarisation Study in Young, Elderly and Type 2 Diabetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: MEC 10-3-050; MET 10-3-050 (Registry Identifier: MET 10-3-050)
Record Dates: First submitted 2011-11-14; First posted 2011-11-22 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Glucose; insulin; Glycocalyx; Muscle; Vascularisation; young; elderly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Neovascularization, Pathologic | interventions — Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glucose drink (Experimental): 75 gram glucose, dissolved in 250 ml water
  Interventions: Dietary Supplement: Glucose
- Placebo (Placebo Comparator): 250 ml water
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Glucose — Glucose drink: 75 gram dextrose monohydrate, dissolved in 250 ml water
  Other Names: GLU
  Arms: Glucose drink
Dietary Supplement: Placebo — 250 ml water
  Other Names: PLA
  Arms: Placebo

SUMMARY:
Aging is accompanied by a progressive loss of skeletal muscle mass and strength, leading to the loss of functional capacity and an increased risk of developing chronic metabolic disease. One of these metabolic diseases interacting with muscle mass is Diabetes Mellitus type 2. Diabetes Mellitus type 2 is characterized by high blood glucose in the context of insulin resistance and relative insulin deficiency. It has become clear that amongst its many actions, insulin is also a vasoactive hormone. Its effect to cause endothelial-nitric oxide dependent vasodilation is physiologic and dose dependent. Recent data suggest that insulin's metabolic and vascular actions are closely linked. This also means that an increase in microvascular perfusion following food intake is more resistant to postprandial insulin release. This physiological process is brought into prominence with increasing age, and even more in type 2 diabetics, and contributes to diminishing glycaemic control. In the present study the investigators will investigate the impact of postprandial insulin release on microvascular recruitment in the oral cavity.

DETAILED DESCRIPTION:
To fulfil the increasing demand for real-time evaluation of micro vascular flow in muscle tissue, new techniques have been evaluated. The conventional systemic hemodynamic and oxygenation parameters are neither specific nor sensitive enough to detect regional perfusion. A more complete evaluation of tissue oxygenation can be achieved by adding noninvasive assessment of perfusion in peripheral tissues to global parameters. Noninvasive monitoring of peripheral perfusion could be a complementary approach that allows very early application throughout the hospital and interventional research. Orthogonal polarization spectral (OPS) is a non invasive technique that uses reflected light to produce real-time images of the microcirculation. The technology has been incorporated into a small hand-held videomicroscope which can be used in both research and clinical settings. OPS can assess tissue perfusion using the functional capillary density (FCD), i.e., the length of perfused capillaries per observation area (measured as cm/cm2).

FCD is a very sensitive parameter for determining the status of nutritive perfusion to the tissue. So far, one of the most easily accessible sites in humans for peripheral perfusion monitoring is the mouth. OPS produces excellent images of the sublingual microcirculation by placing the probe under the tongue. Movement artifacts, semiquantitative measure of perfusion, the presence of various secretions such as saliva and blood, observer-related bias, and malfunction of the apparatus are some of the limitations of the technique.

In the present study we will investigate the impact of postprandial insulin release on microvascular recruitment in the oral cavity.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged between 20-30 or 65-80 years
* BMI < 30 kg/m2
* Non insulin-dependent Diabetes mellitus type 2 patients. Use of oral anti-diabetic agents (TZD's, Metformin and/or a sulfonylurea derivative) is allowed.

Exclusion Criteria:

* Positive history for hypertension
* Smoking
* Hypertension (according to WHO criteria)18
* Use of medication, except for oral blood glucose lowering medication
* All co morbidities interacting with mobility and muscle metabolism of the lower limbs (e.g. arthrosis, arthritis, spasticity/rigidity, all neurological disorders and paralysis).
* HbA1c > 10.0%
* Diagnosed impaired renal or liver function
* Obesity (BMI>30 kg/m2)
* Cardiac disease or cardiovascular problems in history
* Overt diabetic complications

Min Age: 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-10; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Glycocalyx permeability | 30 minutes after ingestion of the drink
  Changes in glycocalyx permeability in young, elderly and type 2 diabetics after ingestion of a glucose or water (placebo) drink. The glycocalyx will be measured during 2 h after ingestion of the drink.

SECONDARY OUTCOMES:
Microvascular density | 3 h after ingestion of glucose drink
  Determination of microvascular density in muscle tissue in young, elderly and type 2 diabetic patients.

CONTACTS AND LOCATIONS:
Overall Officials: LJC van Loon, Professor, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University Medical Center+, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Groen BB, Hamer HM, Snijders T, van Kranenburg J, Frijns D, Vink H, van Loon LJ. Skeletal muscle capillary density and microvascular function are compromised with aging and type 2 diabetes. J Appl Physiol (1985). 2014 Apr 15;116(8):998-1005. doi: 10.1152/japplphysiol.00919.2013. Epub 2014 Feb 27. PMID 24577061